CLINICAL TRIAL: NCT03336814
Title: Evaluation of Early Association of Terlipressin and Norepinephrine During Septic Shock; the TerliNor Study
Acronym: TERLINOR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-07; 2017-000441-43 (EudraCT Number)
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2017-11

CONDITIONS: Septic Shock
Keywords: Terlipressin; norepinephrine
MeSH Terms: conditions — Shock, Septic | interventions — Terlipressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- terlipressin associated with norepinephrine (Experimental)
  Interventions: Drug: Terlipressin
- placebo (physiologic serum) associated with norepinephrine (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Terlipressin — Administration of terlipressine
  Arms: terlipressin associated with norepinephrine
Other: Placebo — Administration of placebo
  Arms: placebo (physiologic serum) associated with norepinephrine

SUMMARY:
In guidelines norepinephrine is the first line vasopressor recommended in case of septic shock. Use of vasopressin is recommended when norepinephrine fails to maintain a mean arterial pressure above 65mmHg or in salvage. Several studies failed to show a superiority of vasopressin over norepinephrine but none evaluated the effect of an early association on organ failure. Terlipressin is a pro-drug of vasopressin which has the same vasoconstrictor effect. We hypothesize that the early association of terlipressin and norepinephrine during septic shock reduces organ failure.

This bi centric, double-blinded, randomised, controlled versus placebo study includes 40 patients. Randomisation will be stratified between centers (two university affiliated intensive care units of Assistance-Publique-Hôpitaux de Marseille, Marseille, France). All patients with septic shock needing more than 0,5µg/kg/min of norepinephrine to reach PAM objectives are randomised, after hemodynamic evaluation and optimisation, to receive continuous infusions of terlipressin (0,01mg/kg/min) or placebo (physiologic serum). The 2 groups receive steroid therapy (continuous intravenous hydrocortisone perfusion) at this time. Clinicians are blinded of perfusion used. Use of terlipressin remains possible in salvage when patients need more of 1µg/kg/min of norepinephrine on physician's decision. Patients with acute ischemic or septic heart failure are excluded of the study.

Primary objective is sepsis related Sequential Organ Failure Assessment (SOFA) score difference between the groups at day 3. Secondary objectives are mortality at day 28, lactates clearance in the first 48hours, renal function (evaluates with AKIN criteria) and use of renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Dose of norepinephrine greater than 0.3 μg / kg / min
* Lactate greater than 2.0 mmol / l

Exclusion Criteria:

* A left heart failure objectified in ultrasound transthoracique by a fraction of left(awkward) ejection of the ventricle lower than 30 % either by thermodilution transpulmonaire with a cardiac index lower than 2,5 l / min / m2 after optimization of the volémie or a central venous saturation in oxygen ( SVcO2) lower than 60 % after optimization of the blood volume.
* Minors
* Pregnant
* Not having terlipressin allergy
* Not having excipient allergy
* A history known for recent acute coronary syndrome (< 3mois)
* An acute coronary syndrome defined by an increase of the troponine and a rise of the segment ST in the electrocardiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-27 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score difference between the groups | Day 3

SECONDARY OUTCOMES:
Mortality rate | Day 28
Lactates clearance | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No